CLINICAL TRIAL: NCT00503308
Title: Patient Perspectives and Testing Uptake With Abbreviated Versus Standard HIV Consenting in the Prenatal Setting: A Randomized-Controlled, Non-Inferiority Trial
Brief Title: HIV Testing Strategies in the Perinatal Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Deborah Cohan, UCSF
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2004-0319
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Results first posted 2011-07-01 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infections; Pregnancy Related
Keywords: HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abbreviated Consenting (Experimental)
  Interventions: Procedure: Abbreviated HIV test counseling
- Standard Consenting (No Intervention)

INTERVENTIONS:
Procedure: Abbreviated HIV test counseling — abbreviated HIV pre-test counseling
  Other Names: opt-out HIV testing
  Arms: Abbreviated Consenting

SUMMARY:
The purpose of the study is to determine whether an abbreviated pretest/post-test CDC recommended counseling is as equally acceptable to prenatal patients as the standard strategy using prenatal care nurses and medical providers at San Francisco General Hospital [SFGH]).

DETAILED DESCRIPTION:
Approximately 40% of HIV-infected infants in the United States in 2000 were born to women not diagnosed with their HIV prior to delivery. (1) There are now effective medical therapies to prevent perinatal transmission, including anti-retroviral therapy, but this requires diagnoses of maternal HIV prior to delivery. Both the Centers for Disease Control and Prevention (CDC) and Institute of Medicine (IOM) have published strong recommendations for universal HIV-antibody testing of pregnant women.

This will be a randomized controlled, non-inferiority trial comparing two HIV testing strategies among English and Spanish-speaking patients presenting for prenatal care at SFGH WHC over the course of approximately one year. Eligible participants will be randomized by study personnel to either standard HIV counseling and testing (control arm) or abbreviated counseling and testing (study arm). Participants will receive a standard prenatal HIV testing brochure, undergo one of two HIV counseling/testing strategies, submit blood for an HIV-1 antibody test, and will follow-up with their medical provider for HIV test results. Upon completion of counseling, participants will undergo a short, structured (Pre-test) questionnaire administered by study staff. Following testing and receipt of results, participants will complete a second (Post-test) structured questionnaire administered by study staff.

Eligible women presenting to SFGH physician or midwife prenatal clinics will be recruited, consented and randomized by study staff to either the standard or abbreviated testing strategy. The outcomes studied will be patient satisfaction and the proportion of study participants who undergo HIV testing. Potential confounder variables to be measured will include demographic characteristics, prior HIV testing history, knowledge about HIV/AIDS, attitudes towards HIV testing, HIV test result, and type of provider (physician versus midwife).

ELIGIBILITY:
Inclusion Criteria:

* Women 16 years of age or above seeking prenatal care at San Francisco General Hospital

Exclusion Criteria:

* Women who do not speak Spanish or English
* Women younger than 16 years of age
* Women who obtained an HIV test during the index pregnancy prior to initiation of prenatal care at SFGH
* Women known to be infected with HIV at initiation of prenatal care at SFGH

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Cohan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Rapid HIV testing of women in labor and delivery: www.cdc.gov/hiv/pubs/rt-women.htm: Centers for Disease Control and Prevention: Divisions of HIV/AIDS Prevention, 2002.
- [Background] Sambamoorthi U, Akincigil A, McSpiritt E, Crystal S. Zidovudine use during pregnancy among HIV-infected women on Medicaid. J Acquir Immune Defic Syndr. 2002 Aug 1;30(4):429-39. doi: 10.1097/00042560-200208010-00009. PMID 12138350
- [Background] Centers for Disease Control and Prevention (CDC). From the Centers for Disease Control and Prevention. Progress toward elimination of perinatal HIV infection--Michigan, 1993-2000. MMWR Morb Mortal Wkly Rep. 2002 Feb 8;51(5):93-7. PMID 11892955
- [Background] Kalish LA, Pitt J, Lew J, Landesman S, Diaz C, Hershow R, Hollinger FB, Pagano M, Smeriglio V, Moye J. Defining the time of fetal or perinatal acquisition of human immunodeficiency virus type 1 infection on the basis of age at first positive culture. Women and Infants Transmission Study (WITS). J Infect Dis. 1997 Mar;175(3):712-5. doi: 10.1093/infdis/175.3.712. PMID 9041351
- [Background] Newell ML. Mechanisms and timing of mother-to-child transmission of HIV-1. AIDS. 1998 May 28;12(8):831-7. doi: 10.1097/00002030-199808000-00004. No abstract available. PMID 9631135
- [Background] Frenkel LM, Cowles MK, Shapiro DE, Melvin AJ, Watts DH, McLellan C, Mohan K, Murante B, Burchett S, Bryson YJ, O'Sullivan MJ, Mitchell C, Landers D. Analysis of the maternal components of the AIDS clinical trial group 076 zidovudine regimen in the prevention of mother-to-infant transmission of human immunodeficiency virus type 1. J Infect Dis. 1997 Apr;175(4):971-4. doi: 10.1086/514003. PMID 9086162
- [Background] Shapiro DE, Tuomala R, Samelson R, et al. Mother-to-Child HIV Transmission Rates According to Antiretroviral Therapy, Mode of Delivery, and Viral Load (PACTG 367): Abstract #114. 9th Conference on Retroviruses and Opportunistic Infections. Seattle, WA, 2002.
- [Background] Phillips KA, Bayer R, Chen JL. New Centers for Disease Control and Prevention's guidelines on HIV counseling and testing for the general population and pregnant women. J Acquir Immune Defic Syndr. 2003 Feb 1;32(2):182-91. doi: 10.1097/00126334-200302010-00010. PMID 12571528
- [Background] Centers for Disease Control and Prevention. Revised recommendations for HIV screening of pregnant women. MMWR Recomm Rep. 2001 Nov 9;50(RR-19):63-85; quiz CE1-19a2-CE6-19a2. PMID 11718473
- [Background] Centers for Disease Control and Prevention (CDC). HIV testing among pregnant women--United States and Canada, 1998-2001. MMWR Morb Mortal Wkly Rep. 2002 Nov 15;51(45):1013-6. PMID 12458916
- [Background] Centers for Disease Control and Prevention (CDC). Advancing HIV prevention: new strategies for a changing epidemic--United States, 2003. MMWR Morb Mortal Wkly Rep. 2003 Apr 18;52(15):329-32. PMID 12733863
- [Background] Ruiz JD, Molitor F, Prussing E, Peck L, Grasso P. Prenatal HIV counseling and testing in California: women's experiences and providers' practices. AIDS Educ Prev. 2002 Jun;14(3):190-5. doi: 10.1521/aeap.14.3.190.23896. PMID 12092921
- [Background] Simpson WM, Johnstone FD, Goldberg DJ, Gormley SM, Hart GJ. Antenatal HIV testing: assessment of a routine voluntary approach. BMJ. 1999 Jun 19;318(7199):1660-1. doi: 10.1136/bmj.318.7199.1660. No abstract available. PMID 10373168
- [Background] Walmsley S. Opt in or opt out: what is optimal for prenatal screening for HIV infection? CMAJ. 2003 Mar 18;168(6):707-8. No abstract available. PMID 12642426
- [Background] Stringer EM, Stringer JS, Cliver SP, Goldenberg RL, Goepfert AR. Evaluation of a new testing policy for human immunodeficiency virus to improve screening rates. Obstet Gynecol. 2001 Dec;98(6):1104-8. doi: 10.1016/s0029-7844(01)01631-3. PMID 11755561
- [Background] Simpson WM, Johnstone FD, Boyd FM, Goldberg DJ, Hart GJ, Prescott RJ. Uptake and acceptability of antenatal HIV testing: randomised controlled trial of different methods of offering the test. BMJ. 1998 Jan 24;316(7127):262-7. doi: 10.1136/bmj.316.7127.262. PMID 9472506
- [Background] Carusi D, Learman LA, Posner SF. Human immunodeficiency virus test refusal in pregnancy: a challenge to voluntary testing. Obstet Gynecol. 1998 Apr;91(4):540-5. doi: 10.1016/s0029-7844(97)00714-x. PMID 9540937
- [Derived] Cohan D, Gomez E, Greenberg M, Washington S, Charlebois ED. Patient perspectives with abbreviated versus standard pre-test HIV counseling in the prenatal setting: a randomized-controlled, non-inferiority trial. PLoS One. 2009;4(4):e5166. doi: 10.1371/journal.pone.0005166. Epub 2009 Apr 15. PMID 19367335

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized-controlled, non-inferiority trial was conducted from October 2006 through February 2008 at San Francisco General Hospital (SFGH), the public teaching hospital of the City and County of San Francisco.
Pre-assignment Details: A total of 278 English- and Spanish-speaking pregnant women were randomized to receive either abbreviated or standard nurse-performed HIV test counseling at the initial prenatal visit.
Groups:
- Standard Consenting Intervention: The standardized HIV pre-test counseling and consent process took approximately 2-5 minutes and reviewed the definition of HIV, modes of transmission and prevention, interpretation of test results and the benefits of testing.
- Abbreviated Consenting Intervention: The intervention arm used a 2-sentence script which lasted approximately 30 seconds.
Period: Overall Study
Arm/Group | Standard Consenting Intervention | Abbreviated Consenting Intervention
Started | 146 | 135
Completed | 144 | 134
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Consenting Intervention | Abbreviated Consenting Intervention | Total
Number analyzed (Participants) | 146 | 135 | 281
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 5 | 13
  Between 18 and 65 years | 138 | 130 | 268
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.99 (6.1) | 26.39 (5.3) | 26.7 (5.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 135 | 281
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 146 | 135 | 281

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With HIV Testing Experience (O'Connor Decisional Conflict Scale)
Description: We measured decisional conflict, the primary outcome of the study, using the English or Spanish language 10-item Low Literacy Decisional Conflict Scale. We considered a DCS score of 25 or less to be low, corresponding to limited conflict. All questions have 3 response categories: yes, no, unsure. Items are scored as 0 = yes, 2 = unsure, 4 = no. Scores for each of the 10 items are summed, divided by 2 and multiplied by 25 to calculate the total score. The final scores range from 0(no decisional conflict) to 100 (extremely high decisional conflict).
Time Frame: same day as HIV test counseling (cross-sectional study)
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Standard Consenting Intervention | Abbreviated Consenting Intervention
Number analyzed (Participants) | 144 | 134
scores on scale | 16.0 [13.1 to 18.9] | 19.9 [16.3 to 23.5]

ADVERSE EVENTS:
Arm/Group | Standard Consenting Intervention | Abbreviated Consenting Intervention
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/135
Other Adverse Events (participants affected / at risk) | 0/146 | 0/135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No